CLINICAL TRIAL: NCT00886964
Title: Immunogenicity and Safety of Intradermal Compare to Intramuscular Hepatitis B Vaccination in HIV Children
Brief Title: Hepatitis B Vaccination (HBV) in HIV Infected Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: ART AIDS Charity Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIV-NAT 107
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: HBV vaccine; HIV children; immune recovery; HBV antibody; Intradermal; Intramuscular; antibody response after HBV vaccine; treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): HBV ID
  Interventions: Biological: Intradermal HBV 1 course
- 2 (Active Comparator): HBV IM
  Interventions: Biological: Intramuscular HBV I course

INTERVENTIONS:
Biological: Intradermal HBV 1 course — Dosage: 2 microgram (mcg), 0.1 ml per dose
  Location: left deltoid area x 1 injection
  Common reactions: local pain, low grade fever, small hyperpigmented induration (granulomatous reaction) which may last up to 6-12 months
  Arms: 1
Biological: Intramuscular HBV I course — Dosage: 2 microgram (mcg), 0.1 ml per dose
  Location: left deltoid area x 1 injection
  Common reactions: local pain, low grade fever, small hyperpigmented induration (granulomatous reaction) which may last up to 6-12 months
  Arms: 2

SUMMARY:
The purpose of this study is :

* To evaluate prevalence of protective hepatitis B antibody comparing intradermal (ID) and intramuscular (IM) route in antiHbsAb negative HIV infected children treated with highly active antiretroviral therapy (HAART)
* To revaccinate the HBV vaccine in the children who didn't have protective HBV Ab

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) and HIV share the same route of transmission and can have co-infection. The prevalence of this co-infection was 8.7% in Thai adult[1, 2] and 12.1% in African HIV vertically transmitted children[3]. Occurrence of HBV has effects to treatment due to having the same medication, lamivudine, tenofovir, emtricitabine or entecavir, to anti HIV medication. HBV can cause chronic liver disease, cirrhosis and hepatocellular carcinoma.

In Thailand, the routine HBV vaccination program was started since 1992. Few reports in severe immune compromise HIV children has been shown to lose their expected preventive measles and hepatitis B antibody from history of scheduled vaccination even after the immune recovery by HAART[4, 5]. Limited data in of prevalence of protective hepatitis B antibody response after immune recovery in Thai HIV infected children treated with highly active antiretroviral therapy. In addition, HBV revaccination in this group of children should be considered[6].

The response of HBV revaccination intramuscularly (IM) at 0, 2 and 6 months in 63 HIV children shown response rates 17.4, 82.5, and 92.1% at 2, 6 and 7 months respectively[6]. Protective anti-HBs were shown in the majority of non-responders to IM HBV vaccine health care workers [21/23 (91.3%)] by two doses of intradermal route (ID)[7].

We hypothesize to see the faster and higher response of antiHBs after first dose of ID compare to IM in anti HBsAb negative HIV infected children. No randomized control trial compare antibody response between IM and ID route in HIV children after immune recovery. The benefit from this trial would be decreased the vaccine cost for resourced limited country.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected individuals
* Age 1-18 years
* Current CD4 within 6 months ≥ 15% or ≥ 200 cells/ml in children age ≥ 6 years
* Signed written informed consent
* Negative HBs Ag, antiHBs, and antiHBc at screening visit

Exclusion Criteria:

* Active AIDS
* Active opportunistic infection
* Platelet < 50,000/ mm3 at screening visit
* History of hypersensitivity to HBV vaccine
* Using oral steroid or immunosuppressive drugs

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2009-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Proportion of children with protective antiHBs at 8 weeks after first dose of HBV ID is superior to HBV IM | 8 weeks

SECONDARY OUTCOMES:
Proportion of children with positive antiHBs at 4 weeks after second and third dose of HBV | 4 weeks
Number of adverse events in HBV ID group and HBV IM group | 7 months
Proportion of protective antiHBs in HIV children after protocol defining immune recovery | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Torsak Bunupuradah, MD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (2):
- Thailand (2):
  - HIV-NAT, Bangkok
  - Pediatric infectious diseases section, King Chulalongkorn Memorial hospital, Bangkok

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org